CLINICAL TRIAL: NCT06929637
Title: The Effect of Amino Acid Infusion on Early Graft Function After Kidney Transplantation
Brief Title: Amino Acid Infusion in Kidney Transplant Recipients
Acronym: AID-KT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, deputy head of Transplant-Nephrology Department, University Hospital, Martin
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TNO_UNM_3
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Short-term Graft Function; Metabolic Effects; Nutritional Effect; Immunological &Amp; Inflammatory Markers; Safety; Adverse Events
Keywords: kidney transplantation; aminoacids; delayed graft function; diabetes mellitus; acute graft rejection; estimated glomerular filtration rate
MeSH Terms: conditions — Delayed Graft Function; Diabetes Mellitus | interventions — Home Infusion Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aminoacid infusion (Active Comparator): Infusion of amino acids,1 g/kg, maximum of 100g AA a day.
  Interventions: Drug: Infusion Therapy
- Placebo arm (Placebo Comparator): Infusion of saline solution
  Interventions: Drug: Saline solution infusion

INTERVENTIONS:
Drug: Infusion Therapy — Infusion of amino acids once daily - dose 1g/kg, maximum 100 g daily for 3 consecutive days starting D1 after kidney transplantation procedure
  Arms: Aminoacid infusion
Drug: Saline solution infusion — Infusion of saline solution a s standard rehydration therapy after kidney transplantation
  Arms: Placebo arm

SUMMARY:
The study addresses the impact of amino acid infusion in the early post-transplant period on graft function and the incidence of post-transplant complications.

DETAILED DESCRIPTION:
Background and Rationale: Delayed graft function (DGF) remains a significant challenge in kidney transplantation, particularly in recipients of deceased donor organs. DGF, often defined as the need for dialysis within the first post-transplant week, is associated with poorer long-term graft survival and increased immunological risk. Ischemia-reperfusion injury (IRI) plays a crucial role in the pathogenesis of DGF, contributing to oxidative stress, inflammation, and endothelial dysfunction. Strategies to mitigate IRI and enhance early graft recovery are highly sought after.

Amino acids play a critical role in cellular metabolism, protein synthesis, and immunomodulation. Prior research suggests that amino acid supplementation may improve nitrogen balance, enhance mitochondrial function, and reduce oxidative stress, potentially benefiting graft recovery. However, there is limited clinical evidence assessing whether perioperative amino acid administration improves graft function in kidney transplant recipients. The AID-KT study aims to evaluate the impact of intravenous amino acid infusion on early graft function following kidney transplantation.

Study Design: AID-KT is a prospective, interventional cohort study with a retrospective control group. The intervention group will receive intravenous amino acid (AA) supplementation at a dose of 1g/kg body weight daily for three days post-transplant. The historical control group consists of kidney transplant recipients from previous years who did not receive amino acid infusion. The study will evaluate graft function, metabolic response, and patient outcomes over a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) undergoing deceased or living donor kidney transplantation
* First-time kidney transplant recipients
* No known allergy or contraindication to amino acids
* Stable hemodynamic status post-transplant
* Signed informed consent

Exclusion Criteria:

* Patients requiring immediate dialysis post-transplant
* Multi-organ transplant recipients
* Severe hepatic dysfunction (Child-Pugh C)
* Uncontrolled infection or sepsis
* Malignancy within the past 5 years (except non-melanoma skin cancer)
* Prior participation in conflicting clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Improving graft function 3 months after kidney transplantation | 90 days after enrollment/kidney transplantation
  Investigators assume infusion of amino acids will improve eGFR in the intervals: 7 days / 14 days / 30 days / 90 days after kidney transplantation.

SECONDARY OUTCOMES:
Decrease of the biopsy proven acute rejection incidence | 90 days after enrollment
  Investigators assume the infusion of amino acids will decrease the incidence of biopsy proven acute rejection in 3rd month after kidney transplantation
Improving levels of total proteins and albumin | 90 days after enrollment/kidney transplantation
  Investigators assume infusion amino acids will improve levels of total proteins and albumin.
Lipid profile improvement | 90 days after enrollment/kidney transplantation
  Investigators assume infusion amino acids will improve levels of total cholesterol, triacyglycerides and LDL-cholesterol.
Decreasing the incidence of delayed graft function | 7 days after enrollment / kidney transplantation
  Investigators assume the infusion of amino acids will decrease the incidence of DGF defined as a need for hemodialysis first week (7 days) after kidney transplantation.
Monitoring the incidence of severe hyperkalemia | 90 days after enrollment/kidney transplantation
  Investigators will compare the safety of infusion if amino acids reflected by the incidence of hyperkalemia > 6.5 mmol/l
Monitoring the incidence of metabolic acidosis | 90 days after enrollment/kidney transplantation
  Investigators will compare the safety of infusion if amino acids reflected by the incidence of metabolic acidosis - serum bicarbonate levels < 20 mmol/l
Monitoring the incidence of elevated liver enzymes | 90 days after enrollment/kidney transplantation
  Investigators will compare the safety of infusion if amino acids with the incidence of increased levels of liver enzymes (AST, ALT, ALP, GMT) > 2x Upper Limit of Normal increased levels of total and conjugated bilirubin > 2x Upper Limit of Normal
Monitoring the incidence of elevated bilirubin | 90 days after enrollment/kidney transplantation
  Investigators will compare the safety of infusion if amino acids with the incidence of increased levels of total and conjugated bilirubin > 2x Upper Limit of Normal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Martin, Martin, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided